CLINICAL TRIAL: NCT02640066
Title: Acupuncture for Acute Viral Lower Respiratory Infection in Hospitalized Children: A Single Blinded Randomized Controlled Trial
Brief Title: Acupuncture for Acute Viral Lower Respiratory Infection in Hospitalized Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 117-15-ZIV
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Viral Respiratory Tract Infection
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental): acupuncture treatment with Supportive care
  Interventions: Other: acupuncture
- standard treatment (No Intervention): Supportive care measures only

INTERVENTIONS:
Other: acupuncture
  Arms: acupuncture

SUMMARY:
Acute viral respiratory infections are among the most common causes of hospitalization in the pediatric population. The usual presentation of viral respiratory tract infections (VRTI) includes fever, malaise, wheezing and or coughing, rhinorrhea and loss of appetite. Up to 50% of children will have at least one viral-induced wheezing illness by school age. Currently treatment of VRTI is essentially supportive and no specific and efficient treatments are known. Given the lack of effective medications, current treatment for severe viral lower respiratory tract infection (LRTI) in infants relies on supportive measures only. These measures include supplementation of oxygen, monitoring of apnea, nasal/gastric tube feeding or intravenous fluids, and, if required, respiratory support with nasal bi-level positive-airway pressure. VTRI therefore represent an important unmet need for improved treatment strategies. Acupuncture's effect on has also been studied. Acupuncture has been shown to be a safe and effective in various respiratory tract inflammations. A review published in 2011 have found that acupuncture is safe for pediatric patients. Acupuncture's effect on acute viral induced wheezing and cough in hospitalized children has yet to be studied. Since the current standard of care is supportive care only, using acupuncture as an additional treatment may provide benefit in reducing wheezing, respiratory distress, and shorten hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* The presence of acute viral respiratory disease

Exclusion Criteria:

* Evidence of chronic cardio-pulmonary disease, immune-suppression or any chronic systemic disease or disability

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
presence of fever | 5 days
presence of cough | 5 days
presence of rhinitis | 5 days
symptoms of pharyngitis | 5 days
presence of crepitations | 5 days
presence of dyspnea or tachypnea | 5 days
  respiratory rate
oxygen saturation | 5 days
  measured by (SpO2)

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel

IPD SHARING:
Plan to Share IPD: No